CLINICAL TRIAL: NCT02998983
Title: Open-label, Multicenter, Phase II Immunotherapy Study With Racotumomab in Patients With High-risk Neuroblastoma
Brief Title: Racotumomab in Patients With High-risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-RACO-2-16
Record Dates: First submitted 2016-12-06; First posted 2016-12-21 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — racotumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Racotumomab (Experimental): Dosage form: intradermal injection. Dosage: 0.4 mg. Frequency: the first 5 doses: biweekly injections; the following 10 doses: monthly injections. Duration: 12 months
  Interventions: Drug: Racotumomab

INTERVENTIONS:
Drug: Racotumomab

SUMMARY:
This clinical trial will be carried out in children diagnosed with high-risk neuroblastoma that have achieved a complete or very good partial response after standard therapy. An additional cohort of children who could not achieve these response criteria or that relapsed after standard therapy but do not have progressive disease will receive Racotumomab together with metronomic chemotherapy.

The main objectives of this study are to determine the immune response after one-year duration immunization with Racotumomab, to describe the response of Racotumomab therapy in minimal residual disease (MRD) in bone marrow and to describe the toxicity profile of Racotumomab.

DETAILED DESCRIPTION:
Neuroblastoma is the most common extra-cranial tumor in childhood but prognosis is still poor, even with the advances in its treatment.

New therapeutic strategies have been examined, and several immunotherapeutic approaches, including combined therapy with monoclonal antibodies (anti-GD2), intravenous interleukin-2 (Il-2) and intravenous granulocyte-macrophage colony-stimulating factor (GM-CSF), and anti-idiotype vaccines are currently being assessed.

Racotumomab is an anti-idiotype antibody capable of inducing anti-N-glycolyl GM3 antibodies in patients with neuroblastoma.

The expression of the ganglioside N-glycolyl GM3 was shown in neuroblastoma and this expression could be useful as a specific target for immunotherapy.

Ractoumomab will be administered once standard therapy for neuroblastoma has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent or written child assent, if applicable, prior to any specific procedure of the study.
2. Aged ≥ 1 year old and ≤ 12 years old at the time of diagnose.
3. High-risk neuroblastoma diagnose according to the International Neuroblastoma Risk Group Staging System (INRGSS) (Annex I).
4. Patients who have received complete chemotherapy, radiotherapy (if applicable) and autologous hematopoietic stem cell transplantation (if applicable) not earlier than 30 days prior to being included in the study, and patients of Group I who have completed therapy with cis retinoic acid or other maintenance onco-specific therapy using the standard dose for neuroblastoma treatment. .
5. Use of concomitant metronomic chemotherapy by patients of Group II is considered acceptable.
6. For patients belonging to other risk group who have relapsed or progressed, the period between the beginning of chemotherapy for the treatment of high-risk neuroblastoma and the inclusion of patients must not exceed 12 months.
7. Partial or complete remission status, very good partial remission or stable disease (pursuant to the International Neuroblastoma Response Criteria) at the time of inclusion (Annex IV).
8. Assessment of the disease must be conducted within 30 days prior to inclusion.
9. Additional studies supporting the response to treatment at the time of inclusion are required.
10. Normal organ functions according to the following parameters:

    * Adequate cardiac function as defined below:
    * Electrocardiogram (ECG) 30 days prior to inclusion without substantial anomalies.
    * Electrocardiogram (ECG) 30 days prior to inclusion with fractional shortening ≥27%
    * Adequate bone marrow functions defined as follows:
    * Neutrophil ≥1000/mm3 with no use of stimulating factor for at least 2 weeks prior to inclusion.
    * Lymphocytes ≥500/mm3
    * Platelets ≥ 50000/mm3.
    * Adequate hepatic functions defined as follows:
    * Direct bilirubin ≤1.5 x upper limit of normal (ULN)
    * AST/ALT ≤ 5 x ULN
    * Adequate renal function defined as follows:
    * Creatinine Clearance ≥70 ml/min/1.73m2 or serum Creatinine (Cr) as per age/gender.
11. Known history of Hepatitis B or C seropositivity with studies showing hepatic function results within acceptable limits may be eligible.
12. Negative HIV serology.
13. Pregnancy test-negative for women of childbearing potential.
14. No previous Racotumomab therapy.
15. No previous intravenous immunoglobulin therapy for at least one month prior to the beginning of treatment.
16. Lansky Scale ≥ 50 (Annex II)
17. Patients with extended bone metastasis in cranial vault or cranial base due to proximity may be considered eligible.

Exclusion Criteria:

In order to be included, patients must not meet the following criteria:

1. Neuroblastoma as progressive disease at the time of the beginning of the study.
2. Patients with known hypersensitivity to any of the components of the investigational drug.
3. Pregnant or breastfeeding patients.
4. Patients who have received other investigational drugs or Racotumomab within 30 days prior to their inclusion in the protocol.
5. History of autoimmune diseases, congenital immunodeficiencies or uncontrolled chronic diseases.
6. Acute allergy disorders or history of severe allergy reactions.
7. History of demyelinating disease or inflammatory disease of the central nervous system or the peripheral nervous system.
8. Patients with any of the following uncontrolled intercurrent disease:

   * Active infectious diseases
   * Uncontrolled cardiac disease: symptomatic congestive heart failure, serious cardiac arrhythmia.
   * Known hepatic disease: cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
   * Convulsions not controlled with any anticonvulsant medication.
9. Other malignancies after adequate therapy showing a disease-free period for more than 5 years.
10. Patients receiving chronic therapy with systemic steroids and other immunosuppressive agents. Topical steroids and inhaled corticosteroids are permitted.
11. History of positive HIV serology.
12. Clinically symptomatic metastasis in central nervous system.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Number of participants who elicit an immune response to a one-year immunization schedule of racotumomab in a cohort study of patients with high-risk neuroblastoma. | 1 year

SECONDARY OUTCOMES:
Number of participants in whom minimally disseminated disease in the bone marrow decreases or disappears with a one-year immunization schedule of racotumomab compared to baseline values at study entry. | 1 year
Number of Participants With Treatment-Related Adverse Events as assessed by CTCAE v4.0 after a one-year immunization schedule of racotumomab when administered alone or together with onco-specific metronomic chemotherapy therapy. | 1 year
Pattern of expression of N-Glycolyl-GM3 gangliosides in tumor samples obtained at disease diagnosis and during follow up if available. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Walter Cacciavillano, MD, Principal Investigator — Prof. Dr. J. P. Garrahan National Children's Hospital
Locations (2):
- Argentina (2):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Prof. Dr. J. P. Garrahan National Children's Hospital, Buenos Aires

IPD SHARING:
Plan to Share IPD: No